CLINICAL TRIAL: NCT03989934
Title: Optimizing a Mindful Intervention for Urban Minority Youth Via Stress Physiology
Brief Title: Teenage Health and Wellness Study
Acronym: THAW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: Johns Hopkins Bloomberg School of Public Health (Other); University of Cincinnati (Other); University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Diana Fishbein, Professor, Department of Human Development and Family Studies, Penn State University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: R61AT009856 (NIH)
Record Dates: First submitted 2019-06-17; First posted 2019-06-18 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Stress; Externalizing Symptoms; Depression Symptoms; Anxiety
Keywords: mindfulness; stress physiology; urban youth
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Mind in Action (Experimental): The Mind in Action is a mindfulness intervention developed by the Holistic Life Foundation (HLF), a Baltimore-based non-profit organization. The curriculum will be delivered over approximately 40 sessions and will follow HLF's typical program modifications for high school students (i.e., sustained focus on breath work and meditation). Each program session will include an initial exercise of focusing on the breath to center oneself, followed by the introduction and practice of different breathing techniques (e.g., rhythmic breathing) that enhance calmness and reduce physiological arousal, and concluding with a brief guided meditation. Instructors will describe benefits of the practices for health and stress management. Participants are given assignments between sessions to reinforce lessons (e.g., breathing exercises or periods of meditation).
  Interventions: Behavioral: The Mind in Action
- Healthy Topics (Active Comparator): Adapted from the Glencoe Health Curriculum (McGraw Hill), Healthy Topics is designed to control for the effects of a positive adult, time and attention, a small group learning environment, engaged instruction, and interesting material. The Healthy Topics curriculum has been successfully implemented as an effective active control condition, with student engagement and participation comparable to the intervention arm. The curriculum includes information about nutrition, exercise, sleep, drug use, and other topics related to physical health.
  Interventions: Behavioral: Healthy Topics

INTERVENTIONS:
Behavioral: The Mind in Action — Mindfulness program for adolescents
  Arms: The Mind in Action
Behavioral: Healthy Topics — Health education program for adolescents
  Arms: Healthy Topics

SUMMARY:
This study evaluates the effects of mindfulness on physiological stress mechanisms implicated in externalizing behaviors and symptoms of affective and traumatic stress among urban adolescents. Program effects on stress physiology will be evaluated using pre- and post-tests of heart rate variability (HRV) during a stress task. Emotional and behavioral outcomes will be measured using student and teacher ratings.

DETAILED DESCRIPTION:
Low-income urban adolescents experience high rates of adversity and trauma exposure, increasing their risk for stress-related problems, including externalizing behaviors and affective and traumatic stress symptoms. These outcomes are associated with dysregulated physiological responses to stress, both in the laboratory and real-world contexts. The neuroplasticity that typifies adolescence heightens vulnerability to stress effects on various brain and body systems. On the other hand, the same neurodevelopmental features also suggest pathways for overcoming and altering stymied trajectories through targeted interventions that leverage the brain's plasticity. Thus, adolescence affords a window of opportunity to reinforce parasympathetic modulation of stress responses, enhancing capacities for emotion regulation and, in effect, protecting against the development of behavioral and affective problems.

There is growing empirical support for the ability of mindfulness-based programs to improve stress management in adults, leading to improved well-being, coping and prosocial behavior. Evidence suggests that mindfulness influences homeostatic systems that modulate neurophysiological responses to stress in the service of emotion regulation. Indeed, neuroimaging studies in adults have established that mindfulness measurably improves brain function, demonstrating the alterability of these mechanisms. No such data have been collected for youth, nor have the psychophysiological mechanisms underlying mindfulness program effects for disadvantaged urban youth been rigorously evaluated. The proposed research thus has potential to substantively advance understanding of mindfulness mechanisms of effects and also to facilitate optimization of mindfulness programming so that it has maximum benefits for urban youth.

This study evaluates the effects of mindfulness on physiological stress mechanisms implicated in externalizing behaviors and symptoms of affective and traumatic stress among urban adolescents. Program effects on stress physiology will be evaluated using pre- and post-tests of heart rate variability (HRV) during a stress task. Emotional and behavioral outcomes will be measured using student and teacher ratings.

ELIGIBILITY:
Inclusion Criteria:

* Must be in the 9th grade at one of the Baltimore City Public Schools participating in the study
* Must provide parental permission and assent.

Exclusion Criteria:

* Students in foster care
* Students in self-contained special education classrooms

Ages: 13 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 203 (Actual)
Dates: Start 2019-02-05 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-06-22 (Actual)

PRIMARY OUTCOMES:
Heart rate variability (HRV) | 25 minutes
  HRV is a biomarker of neural regulation of the autonomic nervous system (ANS) and reflects activity in the parasympathetic (PNS) division. HRV is perturbed by stress and can be altered long-term when adversity is prevalent. As such, it has been associated with symptoms of affective and traumatic stress disorders and externalizing behaviors. We will non-invasively monitor the reactivity of HRV using an earlobe sensor to index the PNS. Participants will complete the Trier Social Stress Task (TSST), which is a standard protocol for inducing moderate psychosocial stress in laboratory settings, and has been widely used with preadolescents and adolescents (Gunnar, Wewerka, Frenn, Long, & Griggs, 2009; Kirschbaum, Pirke, & Hellhammer, 1993). The protocol involves preparing and delivering a speech by the participant in the presence of an adult experimenter and while being videotaped. The trained research assistant is instructed to be as non-responsive as possible during the task.

SECONDARY OUTCOMES:
Child Behavior Checklist: | 10 minutes
  CBCL/4-18 has strong internal consistency and reliability. Considered the standard in field of child psychopathology.
Strengths and Difficulties Questionnaire | 8 minutes
  A 31-item teacher-rated measure assessing aspects of students' social-emotional functioning. We will administer scales for dysregulation and social-emotional competence (13 items total).
Patient-Reported Outcomes Measurement Information System | 6 minutes
  PROMIS is well established and widely used. Includes Depression, Anxiety, Emotional and Behavioral Dyscontrol, Sleep Disturbance, Well Being and Cognitive Function Scales for pediatric samples, from 8-17.
Child PTSD Symptom Scale | 3 minutes
  The CPSS (Foa et al., 2001), which is a 25-item measure of trauma symptoms that has been shown to have good reliability and validity in Baltimore City youth, and has been used in prior studies conducted in Baltimore City public schools.
Emotion Regulation Questionnaire | 3 minutes
  ERQ has 10 items rated on 7-point scale tap individual differences in habitual use of 2 emotion regulation strategies: cognitive reappraisal & expressive suppression (α = .69)
Background Questionnaire | 3 minutes
  Gender, household income, ethnicity/race, mental health treatment received, coping, diet, sleep patterns, etc.
Youth Risk Behavior Survey | 10 minutes
  The YRBS (CDC 2015) includes substance use items, which includes 4 items measuring lifetime use of alcohol, tobacco, and marijuana.
Brief COPE | 5 minutes
  Brief COPE (Carver, 1997), a 28-item measure of various coping skills, including both adaptive and maladaptive coping strategies.
Perceived Stress Scale | 3 minutes
  Perceived Stress Scale: 12 items modified from NIH toolbox (e.g. felt nervous and stressed; able to control irritations). α = 0.89
Child and Adolescent Mindfulness Measure | 3 minutes
  Child and Adolescent Mindfulness Measure (CAMM) (Greco et al., 2011), a brief (10-item) measure of mindfulness that has been found to be reliable and valid in a sample of Baltimore City adolescents. This measure would be given at baseline and post-program, as well as the midpoint of the intervention.
Adverse Childhood Experiences Checklist | 3 minutes
  Adverse Childhood Experiences Checklist (ACEs) (Felitti et al., 1998), a brief (8-item) checklist of trauma exposures adapted from a longer version to exclude items that would require reporting.

CONTACTS AND LOCATIONS:
Overall Officials: Tamar Mendelson, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health; Diana Fishbein, PhD, Principal Investigator — Penn State University
Locations (1):
- Baltimore City Public Schools, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dariotis JK, Mabisi K, Jackson-Gordon R, Rose EJ, Fishbein DH, Mendelson T. Perceived Benefits of Mindfulness and Health Education Programs for Minoritized Adolescents: A Qualitative Analysis. Mindfulness (N Y). 2023 Jun;14(6):1346-1361. doi: 10.1007/s12671-023-02147-y. Epub 2023 Jun 8. PMID 40771868